CLINICAL TRIAL: NCT02564965
Title: Endoscopic Large Caliber Drainage vs. Complete Necrosectomy for Treatment of Walled-off Pancreatic Necrosis: A Prospective, Randomized Noninferiority Trial.
Brief Title: Endoscopic Large Caliber Drainage vs. Complete Necrosectomy for Treatment of Walled-off Pancreatic Necrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-001390
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Necrotizing Pancreatitis
Keywords: Acute Necrotizing Pancreatitis; Walled-Off Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Greater than 50% Necrosis (Other): Subjects who have greater than 50% necrosis as determined by MRI, Endoscopic Ultrasound (EUS), or direct transluminal endoscopic imaging of the collection. This stratification group will be randomized to either the double pigtail plastic stent or the AXIOS metal stent.
  Interventions: Device: Double Pigtail Plastic Stent; Device: AXIOS Metal Stent
- Less than 50% Necrosis (Other): Subjects who have less than 50% necrosis as determined by MRI, Endoscopic Ultrasound (EUS), or direct transluminal endoscopic imaging of the collection. This stratification group will be randomized to either the double pigtail plastic stent or the AXIOS metal stent.
  Interventions: Device: Double Pigtail Plastic Stent; Device: AXIOS Metal Stent

INTERVENTIONS:
Device: Double Pigtail Plastic Stent — Patients will be stratified into two arms (Greater than 50% necrosis or less than 50% necrosis), then will be randomized to either the double pigtail plastic stent or AXIOS metal stent
Device: AXIOS Metal Stent — Patients will be stratified into two arms (Greater than 50% necrosis or less than 50% necrosis), then will be randomized to either the double pigtail plastic stent or AXIOS metal stent
  Other Names: LC-SEMS; Large caliber- self-expanding metal stent

SUMMARY:
The purpose of this study is to determine optimal treatment strategies for symptomatic walled-off pancreatic necrosis( WON).

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 yo) patients
* With symptomatic walled- off pancreatic necrosis in which an endoscopic approach is appropriate based on cross-sectional imaging
* Must have solid necrotic material present in their pancreatic fluid collection as determined by MRI, EUS, or direct transluminal endoscopic imaging of the collection

Exclusion Criteria:

* Previous intervention for pancreatic necrosis (surgical, percutaneous, or endoscopic)
* Indication for emergency laparotomy (compartment syndrome, bowel ischemia, bleeding, or perforation of a GI lumen)
* Uncorrectable coagulopathy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete resolution as defined by complete radiographic resolution of the walled-off necrosis (WON) | Baseline to 4 months after initiation of endoscopic treatment

SECONDARY OUTCOMES:
Clinical resolution of infection as defined by complete radiographic resolution and/or symptoms of pain and gastric outlet obstruction | Baseline to 4 months after initiation of endoscopic treatment
Symptom resolution (Visual Analogue Scale for pain, gastric outlet obstruction, and weight gain) | Baseline to 4 months after initiation of endoscopic treatment
Decrease in incidence of adverse events | Baseline to 4 months after initiation of endoscopic treatment
Decrease in number of hospital days during treatment course | Baseline to 4 months after initiation of endoscopic treatment
Decrease in total costs of pancreatitis-related health care during treatment course | Baseline to 4 months after initiation of endoscopic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Barham Abu Dayyeh, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials